CLINICAL TRIAL: NCT02702960
Title: Sequential, Related Donor Partial Liver Transplantation Followed by Bone Marrow Transplantation for Fibrolamellar or Non-fibrolamellar Hepatocellular Carcinoma (HCC) Including Fibrolamellar HCC
Brief Title: Sequential, Related Donor Partial Liver Transplantation Followed by Bone Marrow Transplantation for Hepatocellular Carcinoma (HCC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was withdrawn due to lack of necessary resources from the liver transplant surgical group.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Fibrolamellar Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J15171; IRB00080373 (Other: JHU IRB)
Record Dates: First submitted 2016-02-26; First posted 2016-03-09 (Estimated); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Fibrolamellar Hepatocellular Carcinoma; Hepatocellular Carcinoma (Fibrolamellar Variant); Hepatocellular Carcinoma
Keywords: FL-HCC; living donor liver transplant; HLA matched first degree relative; Milan Criteria; Ephraim Fuchs; Fibrolamellar Cancer Foundation; fibrolamellar; non-fibrolamellar
MeSH Terms: conditions — Fibrolamellar hepatocellular carcinoma; Carcinoma, Hepatocellular | interventions — Whole-Body Irradiation; Cyclophosphamide; Mesna; Filgrastim; Tacrolimus; Mycophenolic Acid; Prednisone; Antilymphocyte Serum; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- part. liver transplant and BMT (Experimental): Patients receive living related donor partial liver transplantation performed according to standard practices. Patients will be maintained on tacrolimus, MMF, and prednisone after liver transplantation.
  Upon recovery, patient must undergo eligibility screening for bone marrow transplantation (BMT).
  If eligible, patients will begin:
  Antithymocyte globulin (ATG): Day -16 to Day -14; fludarabine: Days -6 to Day -2 low-dose cyclophosphamide: Day -6 and -5. Tacrolimus, mycophenolate mofetil (MMF), and prednisone: day -7 and day -6. Total body irradiation on Day -1 Bone marrow infusion on Day 0. High dose cyclophosphamide plus MESNA: Day 3 and 4th Filgrastim, tacrolimus,MMF, and prednisone: Day 5 until neutrophil counts recover.
  Patients followed up through post transplant day 60, then weekly following discharge.
  Interventions: Procedure: living related donor partial liver transplantation; Radiation: Total body irradiation; Procedure: Bone marrow transplant from same donor; Drug: Cyclophosphamide; Drug: Mesna; Drug: Filgrastim; Drug: Tacrolimus; Drug: mycophenolate mofetil; Drug: Prednisone; Drug: Antithymocyte globulin; Drug: fludarabine

INTERVENTIONS:
Procedure: living related donor partial liver transplantation — HLA matched or haploidentical related living donor partial liver transplant followed by tacrolimus, prednisone, and MMF immunosuppression for >3 wks
Radiation: Total body irradiation — 200 cGy total body irradiation (TBI) on Day -1.
Procedure: Bone marrow transplant from same donor — BMT using cells from the same Human Leukocyte Antigen (HLA)-matched or -haploidentical living related donor will be performed on Day 0
  Other Names: BMT
Drug: Cyclophosphamide — Pre-transplantation low dose cyclophosphamide given day -6 and -5 Post-transplantation high dose cyclophosphamide (PTCy; 50 mg/kg/day) will be administered on Days 3 and 4 with hydration
  Other Names: Cytoxan
Drug: Mesna — administered on Days 3 and 4 with PTCy
  Other Names: sodium-2-mercaptoethane sulfonate
Drug: Filgrastim — administered daily starting on Day 5 until absolute neutrophil count (ANC) recovery
Drug: Tacrolimus — Given after liver transplant for through day -7, stopped on day -6 and restarted on day 5 post BMT
Drug: mycophenolate mofetil — Given after liver transplant for through day -7, stopped on day -6 and restarted on day 5 post BMT
  Other Names: MMF
Drug: Prednisone — Given after liver transplant for through day -7, stopped on day -6 and restarted on day 5 post BMT
Drug: Antithymocyte globulin — Given from Day -16 to Day -14 prior to bone marrow transplantation on day 0
  Other Names: ATG
Drug: fludarabine — fludarabine given from Days -6 to Day -2 before BMT

SUMMARY:
This trial is a phase II, single arm, open-label, single center study to assess a reduced-intensity conditioning regimen, bone marrow transplantation and high dose PTCy in recipients of a partial liver allograft from a Human Leukocyte Antigen (HLA)-matched or -haploidentical living related donor in patients with HCC.

The primary objective of this trial is to characterize recurrence-free survival at 1 year following bone marrow transplantation among recipients of prior partial liver transplantation from the same donor.

DETAILED DESCRIPTION:
The purpose of this study is to characterize the safety and anti-tumor efficacy of sequential partial liver transplantation followed by bone marrow transplantation from the same living related donor. This treatment applies to patients whose cancer remains confined to the liver but is too widespread to be removed by surgery or treated by a liver transplant from a deceased donor. The purpose of this combined treatment is to reduce the risk of the cancer coming back after the liver transplant The bone marrow transplant may reduce the risk of cancer relapse in two ways. First, patients who have combined bone marrow and solid organ transplants may be able to get off all anti-rejection drugs, which inhibit the immune system from destroying cancer cells. Second, the donor's bone marrow contains cells of the immune system, which can attack any cancer cells that remain after the liver transplant.

This trial is a phase II, single arm, open-label, single center pilot study to assess a reduced-intensity conditioning regimen, bone marrow transplantation and high dose post-transplantation cyclophosphamide (PTCy) in recipients of a partial liver allograft from a Human Leukocyte Antigen (HLA)-matched or -haploidentical living related donor in patients with HCC. The trial includes analyses of tumor characteristics and the number and phenotype of tumor infiltrating lymphocytes in the explanted tumor. The trial also includes periodic monitoring of circulating hepatocytes to correlate with tumor response.

The study is expected to take two years to complete accrual of six patients, and the primary objective of this trial is to characterize recurrence-free survival at 1 year following bone marrow transplantation among recipients of prior partial liver transplantation from the same donor. Secondary objectives include documenting percentage of patients who become tolerant of the transplanted liver, i.e. off immunosuppression for >6 months without biochemical evidence of liver rejection, and characterizing the relationship between donor chimerism and transplantation tolerance.

ELIGIBILITY:
Inclusion Criteria:

RECIPIENT

1. Histologic diagnosis of liver-confined fibrolamellar or non-fibrolamellar HCC. Ineligible for curative resection or deceased donor liver transplantation by virtue of NOT meeting the Milan criteria or down-staging criteria:

   1. Single viable tumor ≤5 cm in size or ≤3 tumors each ≤3 cm in size based on CT or Magnetic resonance (MR) imaging
   2. Pretransplant alpha fetoprotein (AFP) level of ≤400.
2. Available human leukocyte antigen (HLA)-matched or -haploidentical, living related donor who is willing to donate bone marrow and part of liver. The donor and recipient must be HLA identical for at least one allele (using high resolution DNA based typing) at the following genetic loci: HLA-A, HLA-B, HLA-C and HLA-DRB1. Fulfilment of this criterion shall be considered sufficient evidence that the donor and recipient share one HLA haplotype.
3. Age 16 to 65 years.
4. Normal estimated left ventricular ejection fraction ( >30% ) and no history of ischemic heart disease requiring revascularization, unless cleared by a cardiologist (as per normal liver and bone marrow (BM) transplant eligibility requirements). Those with an ejection fraction between 30-40%, will require a cardiology consultation and clearance for transplantation.
5. Forced expiratory volume (FEV1) and forced vital capacity (FVC) > 40% of predicted at the screening visit.
6. Serum creatinine <2.0 mg/dl
7. For women of childbearing potential, a negative serum or urine pregnancy test with sensitivity less than 50 milli-International unit (mIU)/m within 72 hours before the start of study medication.
8. Use of two forms of contraception with less than a 5% failure rate or abstinence by all transplanted participants for 12 months after the first dose of study therapy. For the first 60 days post-transplant, recipients should be encouraged to use non-hormonal contraceptives due to the potential adverse effect of hormones on bone marrow engraftment.
9. Ability to receive oral medication.
10. Ability to understand and provide informed consent.
11. Must meet all other criteria for listing for liver transplantation

DONOR:

1. HLA-matched or -haploidentical, parent, child, sibling, or half-sibling of the recipient
2. Meets all requirements for live liver donation based on established criteria
3. Ability to understand and provide informed consent for all study procedures including partial liver transplant and bone marrow harvest.
4. Age < 60 years
5. Body Mass Index (BMI) <35

Exclusion Criteria:

RECIPIENT

1. Extrahepatic disease at the time of enrollment.
2. Macrovascular invasion by tumor as seen on imaging
3. Anti-donor HLA antibody with a level that produces a positive test on flow cytometric crossmatch. [Note: patients with a positive flow cytometric crossmatch may undergo desensitization and may become eligible, at the discretion of the protocol investigators, if desensitization decreases the antibody concentration to a level that produces a negative flow cytometric crossmatch.]
4. Ineligible for liver transplantation per institutional criteria (see Appendix 1)
5. Women who are breastfeeding.
6. History of positive HIV-1 or HIV-2 serologies or nucleic acid test.
7. Active hepatitis B infection as documented by positive Hepatitis B assay
8. Any active, severe local or systemic infection at the screening visit.
9. Use of investigational drug, other than the study medications specified by the protocol, within 30 days of transplantation.
10. Receipt of a live vaccine within 30 days of receipt of study therapy.
11. The presence of any medical condition that the Investigator deems incompatible with participation in the trial.

DONOR

1. Age: less than age 18 or older than age 60
2. BMI >35
3. History of blood product donation to the recipient
4. Significant cardiovascular disease (per cardiology consultation)
5. Significant pulmonary disease (per pulmonology consultation)
6. Significant renal disease
7. History of diabetes mellitus
8. Ongoing malignancies
9. Severe local or systemic infection
10. Severe neurologic deficits
11. Active substance abuse
12. Untreatable/unstable psychiatric illness
13. History of positive HIV-1 or HIV-2 serology or nucleic acid test.
14. Evidence of prior hepatitis B infection as evaluated by hepatitis B surface antigen (HBsAg), total hepatitis B core antibody, and hepatitis B surface antibody (anti-HBsAb).
15. Positive HBV PCR
16. Positive anti-hepatitis C (HCV) antibodies and a positive serum HCV RNA PCR. All positive HCV antibody results must be assessed by an electroimmunoassay enzyme-linked immunosorbent assay (EIA) assay and confirmed by a quantitative serum HCV RNA assay. Participants with positive HCV antibodies but undetectable serum HCV RNA may be considered for eligibility. Participants with negative anti-HCV antibodies but unexplained liver enzyme abnormalities must undergo a quantitative serum RNA assay to rule out false negative HCV serologies.
17. Autoimmune disease requiring immunosuppressive drugs for maintenance.
18. The presence of any medical condition that the Investigator deems incompatible with participation in the trial.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
1 year disease-free survival (at 1 year after BMT) | 1 year
  Disease-free is defined as the lack of radiographic evidence of recurrence by computed tomography or MRI.

SECONDARY OUTCOMES:
Occurrence of Graft versus Host Disease | 1 year
  Determine the cumulative incidences of acute grades II-IV, III-IV and chronic graft-versus-host disease
Death | 1 year
  Proportion of transplanted participants who die
Liver allograft failure | 1 year
  Determine the proportion of transplanted participants with liver allograft rejection demonstrated by a biopsy or clinically if a biopsy cannot be performed.

OTHER OUTCOMES:
Efficacy measure - proportion disease free | 1 year
  The proportion of transplanted participants who remain free of disease recurrence for 1 year post bone marrow transplantation
Efficacy measure- proportion off immunosuppression without graft versus host disease (GVHD) or liver rejection | 1 year
  The proportion of participants who are off immunosuppression without GVHD or liver rejection at 1 year after bone marrow transplantation.

CONTACTS AND LOCATIONS:
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes